CLINICAL TRIAL: NCT07126106
Title: Prospective Validation of the GRADY Bacteremia/Sepsis Prediction Model in Intensive Care Unit Patients: Clinical Performance and Feasibility as an Early Warning System
Brief Title: Prospective Validation of GRADY: A Machine Learning Model for Early Sepsis and Bacteremia Detection in ICU Patients
Status: Recruiting | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, AHMET DOGUKAN, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: dogu-24
Record Dates: First submitted 2025-08-06; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Bacteremia; Sepsis Bacterial
Keywords: Bloodstream Infection; sepsis; Machine Prediction Methods; external validation
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to prospectively validate the GRADY prediction models, which use machine learning algorithms to estimate the risk of gram-negative bacteremia and sepsis in intensive care unit (ICU) patients based on routinely collected vital signs and laboratory data. Sepsis, a life-threatening condition associated with high ICU mortality, requires early diagnosis and treatment-yet current diagnostic methods relying on blood cultures are time-consuming. Existing scoring systems such as SOFA, SIRS, and NEWS2 often lack sufficient sensitivity and specificity in early sepsis detection. Unlike traditional tools, the GRADY models seek to provide earlier and more accurate risk stratification. This study will compare the clinical performance of GRADY models against standard scoring systems and explore their integration as early warning tools to support rapid intervention and improve outcomes in critical care.

DETAILED DESCRIPTION:
Sepsis is a common and critical clinical syndrome encountered in intensive care units (ICUs), associated with high rates of mortality and morbidity. It is defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection (Sepsis-3 definition). Early diagnosis and prompt initiation of appropriate treatment before the onset of organ failure are vital to reducing mortality and morbidity. Gram-negative bacteremia is a significant cause of sepsis cases. Early initiation of appropriate empirical or targeted antibiotic therapy in bacteremia cases plays a pivotal role in patient prognosis. However, the diagnosis of gram-negative bacteremia is generally based on blood culture results, which may take 24-72 hours. The delay during this period is considered a major contributor to increased mortality risk.

In recent years, machine learning-based prediction models have been increasingly used as decision support tools in healthcare. The GRADY prediction models, developed retrospectively in our hospital, aim to predict the risk of sepsis due to gram-negative bacteremia using vital signs and laboratory parameters obtained during routine clinical monitoring. However, prospective validation of these models is essential prior to their integration into clinical practice.

The rationale of this study is to facilitate early identification of ICU patients at risk for bacteremia or sepsis to enable prompt initiation of treatment. Reducing mortality and morbidity through early detection may help alleviate the burden on healthcare systems. Moreover, supporting current clinical practices with early prediction models may enhance decision-making efficiency. The use of early warning systems and machine learning-based algorithms may improve clinical predictive power and allow for timely interventions by clinicians. This study aims to evaluate the diagnostic accuracy and clinical applicability of GRADY models through prospective validation. In this regard, the findings may contribute to the development of new approaches for sepsis and bacteremia management in critical care settings.

In current clinical practice, scoring systems such as the Sequential Organ Failure Assessment (SOFA), Systemic Inflammatory Response Syndrome (SIRS), and National Early Warning Score 2 (NEWS2) are used to define sepsis and to identify high-risk patients early. However, these scoring systems are based on a limited set of clinical and laboratory parameters and have shown suboptimal sensitivity and specificity in early sepsis diagnosis according to various studies. This limitation may reduce the chance of early intervention and negatively affect patient outcomes. GRADY models aim to offer risk prediction based on routinely collected clinical and laboratory data using machine learning algorithms, providing an alternative to conventional scoring systems. This study will compare the diagnostic accuracy and clinical performance of GRADY models with widely used scoring systems such as SOFA, SIRS, and NEWS2.

Currently, there are only a limited number of validated and widely accepted scoring systems available for the early identification of bacteremia. The Pitt Bacteremia Score was developed to predict short-term mortality in patients diagnosed with bacteremia and has been validated in several studies. Unlike the Pitt score, GRADY models aim to predict the risk of bacteremia and sepsis in the early period before diagnosis using routine clinical and laboratory data. Although the two systems do not serve exactly the same purpose, Pitt Bacteremia Scores will be calculated for all patients in this study, and the potential relationship with high-risk classification by the GRADY model will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* ICU stay of 48 hours or longer
* Patients from whom blood cultures were obtained during routine monitoring
* Signed informed consent form

Exclusion Criteria:

* Patients younger than 18 years
* ICU stay shorter than 48 hours
* Patients without blood cultures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who are suspected of having bacteremia while being treated in intensive care will be included in the study.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Gram(-) negative bacteremia | 1-28 days
  Gram (-) bacteria growth in blood culture

SECONDARY OUTCOMES:
SOFA | it will be assessed at the time of patient admission.
  The Sequential Organ Failure Assessment (SOFA) score is a clinical tool that evaluates the extent of a patient's organ dysfunction based on six parameters - respiratory function (PaO₂/FiO₂), coagulation (platelet count), liver function (bilirubin level), cardiovascular status (mean arterial pressure or vasopressor use), central nervous system function (Glasgow Coma Scale), and renal function (creatinine level or urine output) - and it will be assessed at the time of patient admission.
SIRS | they will be assessed at the time of patient admission
  The Systemic Inflammatory Response Syndrome (SIRS) criteria are used to identify a generalized inflammatory state based on four parameters - body temperature, heart rate, respiratory rate or PaCO₂, and white blood cell count
NEWS-2 | it will be assessed at the time of patient admission.
  The National Early Warning Score 2 (NEWS-2) is a clinical scoring system used to assess the severity of a patient's acute illness based on six parameters - respiratory rate, oxygen saturation, systolic blood pressure, heart rate, level of consciousness or new confusion, and temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli etfal research and training hospital, Seyrantepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No